CLINICAL TRIAL: NCT03307187
Title: Group Lifestyle Balance Adapted for Impaired Mobility (GLB-AIM): Translating the GLB to Promote Healthy Weight in People With Mobility Disability (Impairment)
Brief Title: Group Lifestyle Balance Adapted for Individuals With Impaired Mobility (GLB-AIM)
Acronym: GLB-AIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 015-049
Record Dates: First submitted 2017-09-29; First posted 2017-10-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLB-AIM (Experimental): GLB-AIM (Group Lifestyle Balance program, Adapted for individuals with Impaired Mobility) is a 12-month intervention that promotes 5% weight loss by reducing calories and increasing exercise (150 minutes of moderate physical activity). The 23 GLB-AIM sessions were delivered through monthly in-person and teleconference calls and participants were encouraged to self-monitor daily caloric/fat intake and physical activity using materials to accurately measure daily calories and exercise, which included a food scale, measuring cups and spoons and a loaned Garmin vívofit® activity tracker and heart rate monitor. Participants shared their logs with lifestyle coaches over the 13 core sessions and lifestyle coaches provided positive reinforcement, feedback, and problem solving techniques as needed.
  Interventions: Behavioral: GLB Adapted for Individuals with Impaired Mobility
- wait-list control (No Intervention): During the initial 6 month intervention period the control group received several contacts from the study staff via mail that included information on general health (e.g., managing stress, getting good sleep), holiday cards, and scheduling reminders for the 3 and 6 month testing.

INTERVENTIONS:
Behavioral: GLB Adapted for Individuals with Impaired Mobility — The 12-month Group Lifestyle Balance program, Adapted for individuals with Impaired Mobility (GLB-AIM) promotes 5% - 7% weight loss by reducing calories and increasing energy expenditure to 150 minutes of weekly activity. The 23 GLB-AIM sessions were delivered through monthly in-person and teleconference calls. Participants were encouraged to self-monitor daily caloric/fat intake and physical activity using materials to accurately measure daily calories and exercise, which included a food scale, measuring cups and spoons and a loaned Garmin vívofit® activity tracker and heart rate monitor. Participants shared their logs with lifestyle coaches over the 13 core sessions and lifestyle coaches provided positive reinforcement, feedback, and problem solving techniques as needed.
  Arms: GLB-AIM

SUMMARY:
This study tested the effectiveness of the Group Lifestyle Balance™ (GLB) program adapted specifically for people with impaired mobility using standard behavioral approaches for weight loss. The overarching aim of this study was to promote health and reduce chronic disease risk among people with mobility impairment by building an evidence base for weight loss. The central hypothesis was that participants randomized to the intervention arm of the adapted GLB would show significant improvements on primary outcomes of weight and PA compared to a 6-month wait-list control group at 3 and 6 months, and show improvements on several secondary health outcomes.

DETAILED DESCRIPTION:
The following are the specific study aims and hypotheses:

Aim 1: To create an appropriate and usable adaptation of the GLB program for people with mobility impairment.

Hypothesis 1.1: Advisory board participants will identify key adaptations to make the GLB materials appropriate and usable for individuals with impaired mobility.

Aim 2: To establish whether the adapted GLB program for people with mobility impairment is a feasible intervention.

Hypothesis 2.1: Intervention participants will rate the program satisfactorily and attend at least 2/3rd of the weekly group-based meetings and monthly individualized phone calls. Lifestyle coaches will also rate the adapted program satisfactorily.

Aim 3: To determine if the GLB intervention adapted for those with mobility impairment is effective as determined by significant improvement in the primary and secondary outcomes in the intervention group compared to the wait-list control group at 3 and 6 months from baseline.

Hypothesis 3.1: The intervention group will demonstrate significantly greater improvements in our primary outcomes (weight and PA) than the wait list control group at 3 and at 6 months and will show significant improvements in secondary outcomes at 6 months. Hypothesis 3.2: Both groups combined will demonstrate significantly greater improvements in the primary outcomes (weight and PA) after 3, 6 and 12 months of intervention and secondary outcomes after 6 and 12 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years old,
* having a permanent mobility impairment for at least 1 year,
* being overweight as evidenced by BMI > 25 or the equivalent value recommended for spinal cord injury and amputee populations,
* having sufficient upper arm mobility to engage in exercise, having access to a telephone, and
* obtaining physician signed clearance to participate in the weight management intervention.

Exclusion Criteria:

* disabilities for which cognitive impairment substantially impairs autonomy (e.g. mental retardation), as determined by a 5-item everyday autonomy scale,
* medical issues for which exercise is contraindicated such as uncontrolled hypertension or coronary heart disease,
* age 75 or older,
* pregnancy, and
* not fluent in English language.

The upper age cut off is intended to ensure that the sample consists of a population whose permanent mobility impairment is unrelated to aging. Pregnancy is excluded because it is directly related to weight gain.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
weight change | 12 months
  change in weight collected on 4 times over the year. Weight was measured using a Seca accessible scale (#676); wheelchair users were weighed in their chair on the scale, then transferred to a PT mat table from their chair scale to have their chair weighted separately and body weight was calculated as wheelchair weight subtracted from total weight.

SECONDARY OUTCOMES:
Session Attendance | 12 months
  Session attendance recorded for each of the 23 sessions and reported as average attendance at each session
self-monitoring | over 13 core weeks
  self-monitoring adherence for daily food intake
physical activity | baseline, 3, 6, and 12 months
  self reported physical activity reported on the brief International Physical Activity Questionaire as minutes per week spent in moderate-intensity activity, vigorous-intensity activity, moderate and vigorous activity combined, and minutes per week walking/wheeling
waist circumference | baseline, 6, and 12 months
  waist circumference measured while participants laid supine on a PT mat table at the level of the umbilicus, using a fabric measuring tape.
hemoglobin A1c | baseline, 6, and 12 months
  hemoglobin A1c was collected by blood draw and sent to the lab for analysis
blood pressure | baseline, 6, and 12 months
  resting blood pressure after sitting quietly for 10 minutes using an Omron 3 Series wrist worm blood pressure cuff
cholesterol | baseline, 3, 6, and 12 months
  total cholesterol was collected by blood draw during the non-fasting state and sent to the lab for analysis
self-efficacy | baseline, 3, 6, and 12 months
  self-efficacy for health promoting behaviors: 27-items of the Self-Rated Abilities for Health Practices scale which assesses participants perceived ability to engage in health promoting activities across 4 domains (Nutrition, Exercise, Health Practices, Psychological Well Being, plus a total self-efficacy score)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Froehlich Grobe, PhD, Principal Investigator — Baylor Institute for Rehabilitation

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Betts AC, Froehlich-Grobe K. Accessible weight loss: Adapting a lifestyle intervention for adults with impaired mobility. Disabil Health J. 2017 Jan;10(1):139-144. doi: 10.1016/j.dhjo.2016.06.004. Epub 2016 Jun 21. PMID 27431768
- [Derived] Froehlich-Grobe K, Betts AC, Driver SJ, Carlton DN, Lopez AM, Lee J, Kramer MK. Group Lifestyle Balance Adapted for Individuals With Impaired Mobility: Outcomes for 6-Month RCT and Combined Groups at 12 Months. Am J Prev Med. 2020 Dec;59(6):805-817. doi: 10.1016/j.amepre.2020.06.023. Epub 2020 Nov 5. PMID 33160798

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT03307187/Prot_SAP_000.pdf